CLINICAL TRIAL: NCT03715179
Title: Observational Study of Ostomy Consumers
Acronym: OSO
Status: Active, not recruiting | Type: Observational
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 5878-O
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Ostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Ostomates: Individuals living with an ostomy and their caregivers. Participants use their own ostomy pouching systems per their clinician's standard of care

SUMMARY:
The purpose of this longitudinal prospective observational study is to collect electronic Patient Reported Outcome (ePRO) data over a 7-year period directly from people living with an ostomy and their caregivers (participants were re-consented with version 3 of the Protocol in 2020 which indicated a study duration of 5 years, and version 6 of the Protocol in 2025 extending for an additional 2 years). Research participants will be asked to self-report on the ostomy pouching systems they typically use and other various aspects of living with an ostomy and/or caring for an individual living with an ostomy.

DETAILED DESCRIPTION:
This longitudinal prospective observational study is designed as an ePRO registry to collect data from consumers with an ostomy (ileostomy, colostomy, or urostomy) in the United States, Canada, and United Kingdom. An ePRO registry provides a relevant data source founded on the patient's voice. As such, an ePRO registry will be invaluable for prospective observational research aiming to investigate associations of ostomy pouching systems (inclusive of accessories) with peristomal skin health, participant QoL, caregiver burden, product satisfaction, and Healthcare Resource Utilization (HRU). Information from this registry will inform and guide industry healthcare providers and payers in decision-making and subsequent research that factors in the patient and caregiver perspectives. The current study does not test any specific a priori hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age; any self-reported gender
2. Has a single Ileostomy, Colostomy, or Urostomy
3. Is able to provide an informed consent for study participation with no cognitive impairment that would hinder the ability to provide informed consent or provide self-reported data
4. Is willing and able to complete a once per month online questionnaire about life with an ostomy, or has a proxy who can enter data on their behalf
5. Are able to respond themselves or appoint a caregiver as a proxy to respond to online computer questionnaires in English, French Canadian, or Spanish

Caregivers will be entered into this study only if they meet all of the following criteria:

1. Is at least 18 years of age; any self-reported gender
2. Is an informal supporter (such as a relative, friend, or neighbor) of the care recipient
3. Provides support to the care recipient in some capacity (such as ordering supplies or pouch changes) on average at least once per week

Exclusion Criteria:

1. Has more than one stoma
2. Has a single stoma that has been reversed or closed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sponsor-curated customer databases and printed EC/IRB approved advertisements targeted to ostomy product consumers in the United States, Canada, and United Kingdom that may be distributed by clinicians, mail, website, conferences and other consumer contacts.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
To create a patient reported outcomes registry of ostomy consumers | 7 years
  To collect prospective observational data through a patient reported outcome (PRO) registry that will serve as a platform to conduct multiple analyses.

SECONDARY OUTCOMES:
Ostomy specific outcomes | 7 years
  To identify and characterize ostomy specific outcomes for the purposes of hypothesis generation.
Product specific outcomes | 7 years
  To identify and characterize product specific outcomes related to the ostomy specific outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Malandrino, MSN RN CWOCN, Principal Investigator — Hollister Incorporated
Locations (1):
- Hollister Incorporated, Libertyville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colwell JC, Pittman J, Raizman R, Salvadalena G. A Randomized Controlled Trial Determining Variances in Ostomy Skin Conditions and the Economic Impact (ADVOCATE Trial). J Wound Ostomy Continence Nurs. 2018 Jan/Feb;45(1):37-42. doi: 10.1097/WON.0000000000000389. PMID 29300287
- [Background] International Organization for Standardization. ISO 14155:2011: Clinical investigation of medical devices for human subjects - Good clinical practice.
- [Background] ISPE. Guidelines for good pharmacoepidemiology practices (GPP). Pharmacoepidemiol Drug Saf. 2008 Feb;17(2):200-8. doi: 10.1002/pds.1471. No abstract available. PMID 17868186
- [Derived] Scientific and Clinical Abstracts From WOCNext(R) 2022: Fort Worth, Texas diamond June 5-8, 2022. J Wound Ostomy Continence Nurs. 2022 May-Jun 01;49(3 Suppl 1):S1-S99. doi: 10.1097/WON.0000000000000882. No abstract available. PMID 35639023